CLINICAL TRIAL: NCT02378051
Title: Staying Strong With Schools - A School-Based Resilience Support Intervention for Military-Connected Children: A Preliminary Examination of Efficacy
Brief Title: Staying Strong With Schools - A School-Based Resilience Support Intervention for Military-Connected Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Eric Bui, MD, PhD, Eric Bui, MD, PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014P000867
Record Dates: First submitted 2014-09-15; First posted 2015-03-04 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Staying Strong With Schools Intervention; Waitlist Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Staying Strong with Schools Intervention (Experimental): The Staying Strong with Schools Intervention includes: (a) a training of all school professionals, and (b) a year-long training and supervision of the school guidance counselor (RSL), by a Liaison-Trainer (LT).
  Interventions: Behavioral: Staying Strong with Schools Intervention
- Waitlist Control (Placebo Comparator): The waitlist control schools will receive an educational pamphlet outlining resources useful to support military-connected children to be distributed to all educators at the beginning of the Year 1. They will then receive the Staying Strong with Schools Intervention in Year 2.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: Staying Strong with Schools Intervention — 1. On-Site Training to Raise Awareness about the Stress of Parental Deployment and Review Resources Helpful in Promoting military-connected children (MCC)'s Resilience. A 60-minute training will be delivered by our Liaison Trainer on-site to school professionals at the beginning of the school year.
  2. Training and supervision of the Resilience Support Liaison (RSL). In each school receiving the Staying Strong with Schools intervention, we will train the guidance counselor to take on the role of a RSL. The RSL will develop for each MCC an individual resilience support plan that will outline the specific intervention components that will be applied for him/her.
  Arms: Staying Strong with Schools Intervention
Other: Waitlist Control — Receipt of an educational pamphlet outlining resources useful to support military-connected children distributed to all educators at the beginning of the school year.
  Arms: Waitlist Control

SUMMARY:
The purpose of this study is to examine whether Staying Strong With Schools, a school-based intervention to support military-connected children, will be helpful for school professionals and military parents in supporting specific needs of this population of children. As part of the partnership between three school districts in Massachusetts and the Red Sox Foundation and Massachusetts General Hospital Home Base Program, the investigators will examine the efficacy of a training delivered to these schools. The schools will be randomly divided into two groups (like a toss of a coin). Half of the schools will receive the training in 2014-2015, and the other half will be waitlisted and receive the training the following year (2015-2016). All participants (school teachers, military-connected children, and their parents) will be asked to complete questionnaires the first year. The investigators hypothesize that, compared to the control schools, at the end of the school year, SSWS schools will be associated with: (1) greater sense of competence and quality of relationships with military-connected children (MCC) among school professionals; (2) lower parental distress and increased parental sense of competence and general family functioning; and (3) increased social support, and fewer academic, emotional, and behavioral problems among MCC. The investigators hypothesize that an increase in school professionals' sense of competence in identifying and handling MCC's needs, increased quality of relationships with MCC, lower parental distress, increased parental sense of competence, and increased general family functioning will mediate the efficacy of SSWS on MCC's social support and psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

* For school teachers: age 18 or older, employed as teacher in a participating school, willingness to participate in the intervention and able to participate in the informed consent process.
* For military-connected children: age < 18, and currently in grade 1 through 6, student in a participating school, at least one parent who currently serves, or had served in the military since 9/11/01, children without a participating classroom teacher will not receive teacher-rated assessments, but will not be excluded from the school based intervention, parent gives permission for child to participate.
* For military parents: male or female, age 18 or older, parent of a child enrolled in one of the participating schools, parent or co-parent currently serves, or had served in the military since 9/11/01, parent of a military-connected child that is eligible to participate, willing to participate, and able to give informed consent, and permission to release test scores, and have their child participate in SSWS, and self-report, parental and teachers' assessments.

Exclusion Criteria:

* For teachers: unable to attend the initial training, unable to participate in the informed consent process.
* For military-connected children: decline participation, determination by the principal or teacher that participation would not be in the military-connected child's best interest for any reason.
* For military parents: unable to participate in the informed consent process.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The Teachers' Sense of Efficacy Scale | up to two years
  Teachers' Sense of Efficacy is the beliefs in their capability to make a difference in student learning, to be able to get through even to students who are difficult or unmotivated. The Teacher Sense of Efficacy Scale asks teachers to assess their capability concerning instructional strategies, student engagement, and classroom management. It will assess teachers' sense of competence in handling military-connected children's needs.
The Student-Teacher Relationship Scale | up to two years
  The Student-Teacher Relationship Scale (STRS) is widely used to examine teachers' relationships with young students in terms of closeness, conflict, and dependency. It will assess the quality of teachers' relationships with military-connected children.

SECONDARY OUTCOMES:
Parenting Sense of Competence Scale | up to two years
  The Parenting Sense of Competence scale measures parental competence on two dimensions: Satisfaction and Efficacy. It is a 16 item Likert-scale questionnaire (on a 6 point scale ranging from strongly agree [1] to strongly disagree [6]), with nine questions under Satisfaction and seven under Efficacy. Satisfaction section examines the parents' anxiety, motivation and frustration, while the Efficacy section looks at the parents' competence, capability levels, and problem-solving abilities in their parental role.
Depression, Anxiety and Stress Scale | up to two years
  Parental distress will be assessed using the 21-item self-report Depression, Anxiety and Stress Scale. Items each reflect a negative emotional symptom. Each of these is rated on a four-point Likert scale of frequency or severity of the participants' experiences over the last week with the intention of emphasizing states over traits. These scores ranged from 0, meaning that the client believed the item "did not apply to them at all", to 3 meaning that the client considered the item to "apply to them very much, or most of the time".
McMaster Family Assessment Device | up to two years
  Family functioning will be assessed using the general functioning subscale of McMaster Family Assessment Device. The GF subscale consists of 12 questions to permit individuals to rate how well each statement describes their family by selecting among four responses: strongly agree, agree, disagree, strongly disagree.
Behavior Assessment System for Children, Second Edition | up to two years
  Maladaptive and adaptive behaviors and self-perceptions will be assessed using the Behavior Assessment System for Children, Second Edition. In this study, parents will be the informants. This measure assesses child's behaviors in the school setting (Teacher Rating; TRS) as well as the home and community setting (Parent Rating; PRS) without substantial burden.
Child and Adolescent Social Support Scale | up to two years
  Perceived social support will be assessed using the Child and Adolescent Social Support Scale. Subjects respond to items using a six-point scale, ranging from 1= "never," to 6 ="always."

CONTACTS AND LOCATIONS:
Overall Officials: T.H. Eric Bui, MD, PhD, Principal Investigator — Massachusetts General Hospital; Bonnie Ohye, PhD, Principal Investigator — Massachusetts General Hospital
Locations (10):
- United States (10):
  - Community Charter School, Cambridge, Massachusetts
  - East Falmouth Elementary School, East Falmouth, Massachusetts
  - Morse Pond School, Falmouth, Massachusetts
  - Mullen-Hall School, Falmouth, Massachusetts
  - North Falmouth Elementary School, Falmouth, Massachusetts
  - Hyannis West Elementary School, Hyannis, Massachusetts
  - Barnstable United Elementary School, Marstons Mills, Massachusetts
  - West Villages Elementary School, Marstons Mills, Massachusetts
  - Teaticket Elementary School, Teaticket, Massachusetts
  - West Barnstable Elementary School, West Barnstable, Massachusetts